CLINICAL TRIAL: NCT05453877
Title: Clinical Indicators and Brain Image Data: a Cohort Study Based on Kailuan Cohort
Brief Title: Clinical Indicators and Brain Image Data: a Study Based on Kailuan Cohort
Status: Recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: KaiLuan General Hospital (Other)
Responsible Party: Principal Investigator, Wang, Zhenchang, Professor, Beijing Friendship Hospital
Other Study IDs: 202201
Record Dates: First submitted 2022-07-04; First posted 2022-07-12 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Brain Diseases; Hypertension
MeSH Terms: conditions — Brain Diseases; Hypertension

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- subjects from Kailuan community: 1. Age from 18 to 90 years old; 2. Comes from the Kailuan Cohort, completed ≥1 visits which the medical history, physiological indicators were measured; 3. Without contraindications of CT and MR scan; 4. Can cooperate with the measurement of the medical history, physiological indicators and brain imaging.
  Subjects with the following conditions should be excluded:
  1. Known clinical history with congenital or acquired organic diseases (such as aortic stenosis); 2. Known history of drug abuse; 3. Pregnant and lactating women; 4. With clinical history of psychiatric diseases (such as schizophrenia).
  Interventions: Other: No intervention will be applied.

INTERVENTIONS:
Other: No intervention will be applied. — This is an observational study.

SUMMARY:
The investigators will analyze the relationship between the medical history, physiological indicators and the cerebral small vessel disease as well as the structural and functional changes of the brain/head and neck organs in a large sample size of subjects (participants), to identify the influencing factors of the occurrence and development of cerebral small vessel disease as well as the structural and functional changes of the brain/head and neck organs, so as to provide objective clues for early intervention of the disease and improve clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 90 years old;
2. Comes from the Kailuan Cohort, completed ≥1 visits which the medical history, physiological indicators were measured;
3. Without contraindications of CT and MR scan;
4. Can cooperate with the measurement of the medical history, physiological indicators and brain imaging.

Exclusion Criteria:

1. Known clinical history with congenital or acquired organic diseases (such as aortic stenosis);
2. Known history of drug abuse;
3. Pregnant and lactating women; 4. With clinical history of psychiatric diseases (such as schizophrenia).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects from Kailuan Cohorts
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
White matter hyperintensity of the brain measured by MRI (magnetic resonance imaging) | every two years up to 30 years
microbleeds of the brain measured by MRI (magnetic resonance imaging) | every two years up to 30 years
Lacunes of the brain measured by MRI (magnetic resonance imaging) | every two years up to 30 years
Cerebral blood flow measured by MRI (magnetic resonance imaging) | every two years up to 30 years
Brain volume measured by MRI (magnetic resonance imaging) | every two years up to 30 years
White matter microstructural integrity of the brain measured by MRI (magnetic resonance imaging) | every two years up to 30 years

SECONDARY OUTCOMES:
blood glucose level | every two years up to 30 years
Cervical vascular ultrasound | every two years up to 30 years
Fundus color photography of the eyes | every two years up to 30 years
Fundus optical coherence tomography (OCT) | every two years up to 30 years
Blood pressure (both Systolic and Diastolic Blood Pressure) | every two years up to 30 years
BMI (body mass index) | every two years up to 30 years
Uric acid | every two years up to 30 years

OTHER OUTCOMES:
Pulse Wave Velocity, PWV | every two years up to 30 years
Lipoprotein | every two years up to 30 years

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Kailuan General Hospital, Tangshan, Hebei

REFERENCES:
- [Derived] Guo S, Sun J, Zhang Y, Li X, Li J, Zhao X, Zhao P, Chen S, Wu S, Hui Y, Wang Z, Lv H. Association of long-term blood pressure exposure with DTI-ALPS: A population-based cohort study. Brain Res. 2025 Dec 1;1868:149998. doi: 10.1016/j.brainres.2025.149998. Epub 2025 Oct 15. PMID 41106763
- [Derived] Tong N, Hui Y, Gou SP, Chen LX, Wang XH, Chen SH, Li J, Li XS, Wu YT, Wu SL, Wang ZC, Sun J, Lv H. Clinical information prompt-driven retinal fundus image for brain health evaluation. Mil Med Res. 2025 Aug 6;12(1):47. doi: 10.1186/s40779-025-00630-2. PMID 40770361
- [Derived] Zhang T, Lv H, Zhao X, Zeng N, Hui Y, Chen S, Wu N, Xu M, Wu Y, Xing A, Shi H, Zhang S, Liang X, Wang Y, Wu S, Cui L, Wang Z, Liu Y. Serum uric acid is associated with midbrain enlarged perivascular spaces: Results from Multi-modality Medical imaging sTudy bAsed on KaiLuan Study (META-KLS). Prog Neuropsychopharmacol Biol Psychiatry. 2024 Jul 13;133:111000. doi: 10.1016/j.pnpbp.2024.111000. Epub 2024 Apr 3. PMID 38580007
- [Derived] Lv H, Zeng N, Li M, Sun J, Wu N, Xu M, Chen Q, Zhao X, Chen S, Liu W, Li X, Zhao P, Wintermark M, Hui Y, Li J, Wu S, Wang Z. Association between Body Mass Index and Brain Health in Adults: A 16-Year Population-Based Cohort and Mendelian Randomization Study. Health Data Sci. 2024 Mar 15;4:0087. doi: 10.34133/hds.0087. eCollection 2024. PMID 38500551
- [Derived] Sun J, Hui Y, Li J, Zhao X, Chen Q, Li X, Wu N, Xu M, Liu W, Li R, Zhao P, Wu Y, Xing A, Shi H, Zhang S, Liang X, Wang Y, Lv H, Wu S, Wang Z. Protocol for Multi-modality MEdical imaging sTudy bAsed on KaiLuan Study (META-KLS): rationale, design and database building. BMJ Open. 2023 Feb 10;13(2):e067283. doi: 10.1136/bmjopen-2022-067283. PMID 36764715